CLINICAL TRIAL: NCT00115596
Title: Reforming Pediatric Procedural Training: Developing an Evidence-Based Curriculum
Brief Title: Reforming Pediatric Procedural Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Association of Pediatric Program Directors (Other)
Responsible Party: Principal Investigator, Michael Gaies, Instructor in Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CH 05-05-040
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Health Personnel; Healthy
Keywords: Procedure; Training; Simulation; Pediatrics; Curriculum; Evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention Arm (Experimental): 'Formal Curriculum; Low-Fidelity Simulation'
  Residents randomized to the intervention arm will receive the study skills training curriculum (the intervention).
  Interventions: Other: Formal Curriculum; Low-Fidelity Simulation
- Control (No Intervention): Residents randomized to the control arm will receive standard pediatric training.

INTERVENTIONS:
Other: Formal Curriculum; Low-Fidelity Simulation — The intervention was a formal procedural skills training curriculum consisting of didactic lectures and simulation training.
  Arms: Intervention Arm

SUMMARY:
This study is randomized trial of a procedural skills training curriculum utilizing simulation to teach basic procedural skills to pediatric residents.

DETAILED DESCRIPTION:
This study is designed to evaluate a formal curriculum for teaching basic procedures to pediatric interns at Children's Hospital, Boston. The incoming class of interns for the academic year '05-06 will be randomly assigned to participate in the curriculum or not. Four procedures including intravenous catheter insertion, venipuncture (blood drawing), bag-and-mask ventilation, and lumbar puncture (spinal tap) will be taught. Interns will then be tested on their ability to perform these skills on anatomic models and on live patients. Our hypothesis is that interns receiving the formal curriculum will be more confident and more successful in performing these procedures than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Intern in the Boston Combined Residency Program for AY '05-'06

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
1. Percent successful IV placement over 6 months | 6/19/2005 - 6/30/2006
  % IVs successfully placed
2. Percent successful venipunctures over 6 months | 6/19/2005 - 6/30/2006
  % venipunctures with adequate sample for testing
3. Score on lumbar puncture subcomponent checklist on simulator at 6 months | 6/19/2005 - 6/30/2006
  % steps correct on checklist
Score on bag mask ventilation 9BMV) subcomponent checklist on simulator at 6 months. | 6/19/2005 - 6/30/2006
  % steps correct on checklist

SECONDARY OUTCOMES:
Bag Mask Ventilation: 1. Percentage able to successfully ventilate simulator at 0 and 6 months | 6/19/2005 - 6/30/2006
  Percentage able to successfully ventilate simulator at 0 and 6 months
Average score on BMV checklist at 6 months | 6/19/2005 - 6/30/2006
  Average score on subcomponent checklist at 6 months
Average time to success at 0 and 6 months | 6/19/2005 - 6/30/2006
  Average time to success at 0 and 6 months
4. Score (%) on BMV written test at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score (%) on written test at 0 and 6 months
5. Average likert scale scores on confidence with BMV at 6 months | 6/19/2005 - 6/30/2006
  Average likert scale scores on confidence with procedures at 6 months
IV insertion: 1. Percent successful PIV insertion on simulator at 0 and 6 months | 6/19/2005 - 6/30/2006
  Percent successful PIV insertion on simulator at 0 and 6 months
Score (%) on PIV subcomponent checklist at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score (%) on subcomponent checklist at 0 and 6 months
Score (%) on PIV written test at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score on written test
Average likert scale scores on confidence with PIV at 6 months | 6/19/2005 - 6/30/2006
  Likert scale score
Venipuncture: 1. Percent successful VP insertion on simulator at 0 and 6 months | 6/19/2005 - 6/30/2006
  % VP successul on simulator
2. Score (%) on VP subcomponent checklist at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score on checklist
3. Score (%) on VP written test at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score on written test
4. Average likert scale scores on confidence with VP at 6 months | 6/19/2005 - 6/30/2006
  Likert score
Lumbar puncture: 1. Percentage of atraumatic LP attempts over 6 months | 6/19/2005 - 6/30/2006
  Successful LPs on patients
2. Score (%) on LP subcomponent checklist on simulator at 6 months | 6/19/2005 - 6/30/2006
  Score on checklist
3. Score (%) on subcomponent checklist on first live patient LP | 6/19/2005 - 6/30/2006
  checklist score
4. Number of LP attempts needed to demonstrate competence | 6/19/2005 - 6/30/2006
  number of LPs
5. Score (%) on LP written test at 0 and 6 months | 6/19/2005 - 6/30/2006
  Score on written test
6. Average likert scale scores on confidence with LP at 6 months | 6/19/2005 - 6/30/2006
  Likert score

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Gaies, MD MPH, Principal Investigator — Childrens's Hospital, Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States